CLINICAL TRIAL: NCT05907291
Title: A 12-week, Phase 2 Open-label, Sequential Dose Cohort Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of CRN04894 Treatment in Participants With Congenital Adrenal Hyperplasia (TouCAHn)
Brief Title: Evaluate the Safety, Efficacy, and Pharmacokinetics of CRN04894 in Participants With Congenital Adrenal Hyperplasia (TouCAHn)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRN04894-03; 2023-503488-40-00 (Other: European Medicines Agency)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Congenital Adrenal Hyperplasia; Classic Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; CAH; TouCAHn; CRN04894; atumelnant
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential Dose (Experimental): Sequential, open-label, 12-week fixed-dose cohorts.
  Interventions: Drug: atumelnant (CRN04894)

INTERVENTIONS:
Drug: atumelnant (CRN04894) — Atumelnant is an orally active nonpeptide melanocortin 2 receptor (MC2R) or adrenocorticotropic hormone (ACTH) antagonist.

SUMMARY:
The purpose of this Phase 2, open-label, sequential dose cohort study is to evaluate the safety, efficacy, and pharmacokinetics (PK) of atumelnant (CRN04894) in participants with classic congenital adrenal hyperplasia (CAH) caused by 21-hydroxylase deficiency.

DETAILED DESCRIPTION:
This Phase 2, open-label, sequential dose cohort study will evaluate the efficacy, safety, PK, and PD of atumelnant (CRN04894) when administered for 12 weeks in participants with CAH caused by 21-hydroxylase deficiency. Up to 42 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 to 75 years of age at the time of signing the Informed Consent Form (ICF). Participants ≥16 years of age may be included in sites located in the United States
2. Classic 21-hydroxylase deficiency
3. On a stable regimen of glucocorticoid replacement (eg, hydrocortisone, prednisolone, prednisone, methylprednisolone)
4. Compliance with glucocorticoid replacement and mineralocorticoid replacement (if applicable) regimen during the Screening Period
5. Minimum total daily dose of ≥15 mg hydrocortisone (or equivalent). For Cohort 4, a mean daily dose of ≥11 mg/m²/day of hydrocortisone or hydrocortisone equivalents will be used for inclusion
6. If on estrogen therapy (any route), dose must be stable for at least 3 months prior to Screening

Exclusion Criteria:

1. Diagnosis of any other form of CAH other than classic 21-hydroxylase deficiency
2. Dexamethasone use within 30 days of Screening for Cohorts 1-3. In Cohort 4, dexamethasone is permitted
3. History of bilateral adrenalectomy, hypopituitarism, or other condition requiring chronic glucocorticoid therapy
4. Night shift workers or any other reason for abnormal sleep/wake cycles
5. Clinically significant unstable medical condition or chronic disease other than CAH
6. History of major surgery/surgical therapy for any cause within 4 weeks prior to Screening
7. Diabetes mellitus treated with insulin for less than 6 weeks prior to Screening, or with change in total daily insulin dose by >15% within 6 weeks prior to Screening
8. Poorly controlled diabetes mellitus defined as having a hemoglobin A1c (HbA1c) ≥8.5%(≥69 mmol/mL), or estimated HbA1c based on fructosamine if HbA1c is not evaluable (eg, due to hemoglobinopathies)
9. Participants with hypothyroidism who are not receiving adequate hormone replacement therapy based on thyroid hormone levels measured at the time of Screening
10. History of unstable angina or acute myocardial infarction within 12 weeks prior to Screening or other clinically significant cardiac disease at the time of Screening
11. History of cancer excluding cured/treated dermal squamous or basal cell carcinoma or cervical carcinoma in situ
12. Pregnant or lactating
13. Known history of illicit drug or alcohol abuse within the last year
14. Use of antiandrogen therapy in the past 3 months (eg, spironolactone, finasteride, cyproterone acetate, flutamide)
15. Use of testosterone, androgen-containing supplements, aromatase inhibitors, or growth hormone

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in morning (before 11:00) serum androstenedione (A4) | Week 12
Incidence of treatment-emergent adverse events (TEAEs) throughout the study | Week 12

SECONDARY OUTCOMES:
Change from baseline in morning (before 11:00) serum 17-hydroxyprogesterone (17-OHP) | Week 12

CONTACTS AND LOCATIONS:
Locations (26):
- United States (8):
  - Crinetics Study Site, Pasadena, California
  - Crinetics Study Site, Ann Arbor, Michigan
  - Crinetics Study Site, Minneapolis, Minnesota
  - Crinetics Study Site, St Louis, Missouri
  - Crinetics Study Site, Morehead City, North Carolina
  - Crinetics Study Site, Cleveland, Ohio
  - Crinetics Study Site, Philadelphia, Pennsylvania
  - Crinetics Study Site, East Providence, Rhode Island
- Argentina (2):
  - Crinetics Study Site, Córdoba, Córdoba Province
  - Crinetics Study Site, Buenos Aires
- Brazil (7):
  - Crinetics Study Site, Curitiba, Paraná
  - Crinetics Study Site, Rio de Janeiro, Rio de Janeiro
  - Crinetics Study Site, Porto Alegre, Rio Grande do Sul
  - Crinetics Study Site, Botucatu, São Paulo
  - Crinetics Study Site, Ribeirão Preto, São Paulo
  - Crinetics Study Site, São Paulo, São Paulo
  - Crinetics Study Site, São Paulo
- Crinetics Study Site, Munich, Bavaria, Germany
- India (2):
  - Crinetics Study Site, Bangalore, Karnataka
  - Crinetics Study Site, Vellore, Tamil Nadu
- Italy (3):
  - Crinetics Study Site, Napoli
  - Crinetics Study Site, Roma
  - Crinetics Study Site, Rozzano
- United Kingdom (3):
  - Crinetics Study Site, Sheffield, South Yorkshire
  - Crinetics Study Site, Coventry, West Midlands
  - Crinetics Study Site, London

IPD SHARING:
Plan to Share IPD: No